CLINICAL TRIAL: NCT01764152
Title: Efficiency in Population of Influenza Vaccination for Seasonal 2012-2013 for Flu Prevention of the Hospitalized Adults: an Observational Study
Brief Title: Clinical Trial to Assess the Influenza Vaccination (FLUVAC 02)
Acronym: FLUVAC EV-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C12-57; 2012-A01118-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-12-21; First posted 2013-01-09 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-03

CONDITIONS: Adult Hospitalized
Keywords: Prevention,; influenza,; adults hospitalized,; vaccines,; Effectiveness
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasopharyngeal sample (Experimental): one will be taken nasopharyngeal all patients hospitalized for 24 hours with ILI in the last seven days.
  Interventions: Other: nasopharyngeal sample

INTERVENTIONS:
Other: nasopharyngeal sample — The nasopharyngeal sample will be used to find the types and subtypes of influenza virus and other respiratory viruses.

SUMMARY:
This study assesses the seasonal of influenza vaccine effectiveness in adults hospitalised with laboratory-confirmed influenza through a network of hospitals in France

DETAILED DESCRIPTION:
Influenza vaccination strategies aim at protecting high-risk population from severe outcomes. Estimating the effectiveness of seasonal vaccines against influenza related hospitalisation is important to guide these strategies. The objective is to measure the population effectiveness of influenza vaccine in patients hospitalized with virologically confirmed influenza laboratory during the influenza season 2012/2013 in a French hospitals network. This is a study "case-control" involving a nasopharyngeal sample for all hospitalised patients presenting an influenza-like illness within seven days. Cases will be patients RT-PCR positive for influenza. Controls will be patients negative for any influenza virus.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Affiliated with social security health insurance
* Written informed consent
* Patients hospitalized for 24 hours and presenting an influenza-like illness in the last 7 days before the hospitalization

Exclusion Criteria:

* Against indication for influenza vaccination(Hypersensitivity to the active substances, to any of the excipients and to trace eg eggs, including ovalbumin, chicken protein)
* Patients institutionalized without regular community interaction
* Patient already hospitalized for respiratory infection during the 2012-2013 influenza season
* Flu already virologically documented in the current influenza season 2012-2013 (RT-PCR, multiple RT-PCR and / or culture.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Measure of vaccine efficacy in population by comparing the number of influenza cases virologically documented in hospitalized patients vaccinated and unvaccinated. | 6 months
  The effectiveness of the vaccine in population will be calculated according to the formula VE = 1 - OR. an interval exact confidence of 95% will be calculated on the point estimate.

SECONDARY OUTCOMES:
Measure of vaccine efficacy in population by comparing the number of influenza cases virologically documented in hospitalized patients vaccinated and unvaccinated according to age groups | 6 months
Measure of vaccine efficacy in population by comparing the number of influenza cases virologically documented in hospitalized patients vaccinated and unvaccinated depending on the subtypes. | 6 months
Description of the population hospitalized for ILI (socio-demographic characteristics, risk factors, pattern and duration of hospitalization...) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Institut National de la Santé Et de la Recherche Médicale, Paris, France

REFERENCES:
- [Background] Puig-Barbera J, Tormos A, Sominina A, Burtseva E, Launay O, Ciblak MA, Natividad-Sancho A, Buigues-Vila A, Martinez-Ubeda S, Mahe C; GIHSN Group. First-year results of the Global Influenza Hospital Surveillance Network: 2012-2013 Northern hemisphere influenza season. BMC Public Health. 2014 Jun 5;14:564. doi: 10.1186/1471-2458-14-564. PMID 24903737
- [Background] Puig-Barbera J, Natividad-Sancho A, Launay O, Burtseva E, Ciblak MA, Tormos A, Buigues-Vila A, Martinez-Ubeda S, Sominina A; GIHSN Group. 2012-2013 Seasonal influenza vaccine effectiveness against influenza hospitalizations: results from the global influenza hospital surveillance network. PLoS One. 2014 Jun 19;9(6):e100497. doi: 10.1371/journal.pone.0100497. eCollection 2014. PMID 24945510